CLINICAL TRIAL: NCT00593736
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel, Proof of Concept Study to Evaluate the Effectiveness of Ramelteon to Advance the Timing of Sleep in Individuals With Delayed Sleep Phase Syndrome (DSPS)
Brief Title: Efficacy of Ramelteon on Speeding Up Sleep in Subjects With Delayed Sleep Phase Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-04-TL-375-044
Record Dates: First submitted 2008-01-02; First posted 2008-01-15 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Sleep Disorders, Circadian Rhythm
Keywords: Delayed sleep phase syndrome; drug therapy
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm | interventions — ramelteon

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ramelteon 1 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 4 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Ramelteon 8 mg QD (Experimental)
  Interventions: Drug: Ramelteon
- Placebo QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ramelteon — Ramelteon 1 mg, tablets, orally, once daily for up to two weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 1 mg QD
Drug: Ramelteon — Ramelteon 4 mg, tablets, orally, once daily for up to two weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 4 mg QD
Drug: Ramelteon — Ramelteon 8 mg, tablets, orally, once daily for up to two weeks.
  Other Names: Rozerem™; TAK-375
  Arms: Ramelteon 8 mg QD
Drug: Placebo — Ramelteon placebo-matching tablets, orally, once daily for up to two weeks.
  Arms: Placebo QD

SUMMARY:
The purpose of this study is to evaluate the ability of ramelteon, once daily (QD), to advance the timing of sleep in individuals with delayed sleep phase syndrome.

DETAILED DESCRIPTION:
Delayed sleep phase syndrome is the most common circadian disorder in adolescents and most adults with the condition report onset of symptoms during childhood or adolescence. Delayed Sleep Phase Syndrome involves a chronic mismatch between the usual daily schedule required by the individual's environment and his or her circadian sleep wake pattern. Individuals suffering from delayed Sleep Phase Syndrome experience great difficulty when attempting to fall asleep before 1-2 am, if not later, as well as rising at acceptable hours of the morning despite having completely normal sleep architecture and sleep duration. Delayed Sleep Phase Syndrome is a sleep disorder that results from a dysregulation of the circadian sleep-wake rhythm. Delayed Sleep Phase Syndrome is often the cause of severe insomnia and is associated with excessive daytime sleepiness, major depressive disorder and severe disruption of education, work and social functioning. Its major symptom is extreme difficulty initiating sleep at a conventional hour and waking on time in the morning for school or work.

Ramelteon is a selective melatonin type 1 (MT1) and type 2 (MT2) receptor agonist. The purpose of this study is to evaluate the ability of ramelteon to advance the timing of sleep in individuals with delayed sleep phase syndrome. The effect of ramelteon will be analyzed based on collection of information from a post-sleep questionnaire completed by participants, and data collected by polysomnography in a sleep clinic setting. Total participation time involved in this study will be approximately 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females of childbearing potential who is sexually active must agree to use adequate contraception from screening throughout the duration of the study.
* Must have a diagnosis of Delayed Sleep Phase Syndrome according to International Classification of Sleep Disorders criteria for at least 3 months.
* Based on sleep history, subject's habitual sleep time is more than 3 hours later than the desired sleep time.
* Must have had self reported insomnia which is defined per the sleep history as his or her sleep latency of at least 45 minutes when attempting to sleep at desired sleep time required by his or her work or school schedule.
* The subjective sleep latency via Post sleep questionnaire during outpatient screening period must be greater than or equal to 45 minutes during every working night or school night provided the subject went to bed at their desired sleep time.
* During single blind placebo run-in Polysomnography screening nights, subject is instructed to go to bed at their desired bed time and must demonstrate difficulty in falling asleep based on the following criteria:

  * During Polysomnography screening nights when the subject goes to bed at their desired sleep time or
  * The average of total wake time
* Is in good health as determined by a medical and psychiatric history, physical examination, Electrocardiogram, and serum chemistry and hematology.
* Is able to complete self-rating scales via interactive voice response system, and has a touch tone phone.
* Is willing to comply with study procedures and restrictions with fixed sleep time and wake time during the study and to attend regularly scheduled clinic visits as specified in this protocol.
* Has a body mass index is between 18 and 34 kg/m2, inclusive.
* Has a negative urine test result for selected substances of abuse (including alcohol).
* Has a negative test result for hepatitis B surface antigen and hepatitis C virus antibody or history of human immunodeficiency virus.
* Has not used pharmacological sleep assistance for more than 4 times/week during the 3 months prior to Initial Screening.
* Must have discontinued use of all pharmacological sleep aids beginning 1 week prior to Visit 2 and for the duration of the trial.

Exclusion Criteria:

* Has a known hypersensitivity to ramelteon or related compounds, including melatonin and melatonin-related compounds or 5-hydroxytryptophan.
* Has participated in any other investigational study and/or taken any investigational drug within 30 days or 5 half-lives prior to the first dose of study medication, whichever is longer.
* Has flown across greater than 3 time zones within the past 3 months prior to administration of study medication.
* Has sleep schedule changes required by employment (eg, shift worker) within 3 months prior to the administration of study medication.
* Has participated in a weight loss program or has substantially altered their exercise routine within 30 days prior to the administration of study medication.
* Has a history of alcohol abuse within the past 12 months, as defined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision, or regularly consumes more than 14 alcoholic drinks per week or consumes any alcoholic drinks within 24 hours of Screening Visit.
* Has a history of drug abuse within the past 12 months.
* Has a current, clinically significant neurological (including cognitive), hepatic, renal, endocrine, cardiovascular, gastrointestinal, pulmonary, hematological, or metabolic disease, as determined by the investigator.
* Has a probable current diagnosis of another circadian rhythm disorder or a sleep disorder other than Delayed Sleep Phase Syndrome that is the primary cause of insomnia.
* Had an apnea hypopnea index greater than 10 on the first night of Polysomnography Screening.
* Has periodic limb movements during sleep with arousal index greater than 10 as seen on the first night of Polysomnography screening only.
* Has a positive urine drug screen or breathalyzer test.
* Has ever had a history of seizures; sleep apnea, restless leg syndrome, chronic obstructive pulmonary disease, fibromyalgia, or a positive test result for the aforementioned ailments on the screening Polysomnography, schizophrenia, bipolar disorder, mental retardation, or cognitive disorder.
* Has a history of psychiatric disorder (including anxiety or depression) within the past 12 months.
* Smokes more than 3 cigarettes per day or uses tobacco products during nightly awakenings.
* Routinely consumes caffeine including coffee, tea and/or other caffeine-containing beverages or food averaging more than 600 mg of caffeine per day.
* Has used any central nervous system drug or other medications, including those used to treat psychiatric disorders, known to affect sleep/wake function within 1 week whichever is longer prior to the administration of single blind study drug.
* Used melatonin, or other drugs/supplements known to affect sleep/wake function within 1 week (or 5 half lives of the drug) whichever is longer prior to the first dose of single blind medication.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Anxiolytics
  * Hypnotics
  * Antidepressants
  * Anticonvulsants
  * Sedating H1 antihistamines
  * Systemic steroids
  * Respiratory stimulants
  * Decongestants
  * Antipsychotics
  * Muscle relaxants
  * Over-the-counter and prescription diet aids
  * Narcotic analgesics
  * Beta Blockers
  * St. John's wort
  * Kava kava
  * Ginkgo biloba
  * Modafinil
  * Coumadin
  * Heparin
  * Melatonin and all other drugs or supplements known to affect sleep/wake function will be prohibited within 1 week of the first dose of study medication and during the entire study.
* Has any clinically important abnormal finding as determined by a medical history, physical examination, Electrocardiogram, or clinical laboratory tests as determined by the investigator.
* Has a positive hepatitis panel including anti- Hepatitis A Virus, hepatitis B surface antigen or anti- hepatitis C virus.
* Has any additional condition(s) that in the investigator's opinion would:

  * Affect sleep/wake function
  * Prohibit the subject from completing the study, or
  * Not be in the best interest of the subject.
* Exhibits a placebo response during single-blinded placebo run in period.
* Individuals with a habitual sleep time later than 4:00 am should not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2007-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (42):
- United States (42):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Fountain Valley, California
  - Glendale, California
  - Los Angeles, California
  - San Diego, California
  - Santa Monica, California
  - Tustin, California
  - Colorado Springs, Colorado
  - Hallandale Bch, Florida
  - Naples, Florida
  - Pembroke Pines, Florida
  - South Miami, Florida
  - Spring Hill, Florida
  - St. Petersburg, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Gainesville, Georgia
  - Macon, Georgia
  - Chicago, Illinois
  - Danville, Indiana
  - Overland Park, Kansas
  - Topeka, Kansas
  - Crestview Hills, Kentucky
  - Paducah, Kentucky
  - Chevy Chase, Maryland
  - Newton, Massachusetts
  - Hattiesburg, Mississippi
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - New York, New York
  - Raleigh, North Carolina
  - Salisbury, North Carolina
  - Cincinnati, Ohio
  - Dublin, Ohio
  - Toledo, Ohio
  - Salem, Oregon
  - Clarks Summit, Pennsylvania
  - Columbia, South Carolina
  - Austin, Texas

REFERENCES:
- See also: Rozerem Package Insert — http://general.takedapharm.com/content/file/pi.pdf?applicationcode=ab2d7112-8eb3-465a-8fda-35018a9eafb0&fileTypeCode=ROZEREMPI

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects enrolled at 47 sites in the United States from 10 October 2007 to 23 May 2008.
Pre-assignment Details: Subjects were screened for 14 days, entered a 7-day placebo run-in, and then were randomized to once-daily (QD) treatment. To enter the double-blind randomization period, subjects must have met the eligible inclusion and none of the exclusion criteria and met sleep diagnostic criteria established during screening polysomnography.
Groups:
- Ramelteon 1 mg QD: Ramelteon 1 mg, tablets, orally, once daily for up to 2 weeks.
- Ramelteon 4 mg QD: Ramelteon 4 mg, tablets, orally, once daily for up to 2 weeks.
- Ramelteon 8 mg QD: Ramelteon 8 mg, tablets, orally, once daily for up to 2 weeks.
- Placebo QD: Ramelteon placebo-matching tablets, orally, once daily for up to 2 weeks.
Period: Screening Period and Placebo Run-in
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Started | 0 | 0 | 0 | 549
Completed | 0 | 0 | 0 | 132
Not Completed | 0 | 0 | 0 | 417
Not completed — Adverse Event | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 9
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 43
Not completed — Study Termination | 0 | 0 | 0 | 15
Not completed — Did Not Meet Criteria | 0 | 0 | 0 | 322
Not completed — Various | 0 | 0 | 0 | 25
Period: Treatment Period and Placebo Run-out
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Started | 32 | 33 | 35 | 32
Completed | 29 | 31 | 30 | 28
Not Completed | 3 | 2 | 5 | 4
Not completed — Lost to Follow-up | 2 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 3
Not completed — Various | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD | Total
Number analyzed (Participants) | 32 | 33 | 35 | 32 | 132
Age Continuous [Mean (Standard Deviation); unit: years] | 29.6 (9.36) | 33.7 (12.31) | 29.3 (9.40) | 33.1 (13.08) | 31.4 (11.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 17 | 12 | 64
  Male | 14 | 16 | 18 | 20 | 68
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 19 | 19 | 18 | 75
  Not Hispanic or Latino | 13 | 14 | 16 | 14 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1
  Black or African American | 4 | 3 | 3 | 3 | 13
  White | 24 | 30 | 32 | 28 | 114
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Pharmacologic sleep aid needed to sleep [Number; unit: subjects] — For the question, "Do you use of pharmacological assistance to sleep," an answer of 'no'=0 and 'yes' resulted in the question, "If yes, how often per week?" 1=1 day/week; 2=2 days/week; 3=3 days/week; 4=4 days/week; >4=more than 4 days/week.
  subjects
    0 | 31 | 30 | 33 | 32 | 126
    1 | 0 | 0 | 1 | 0 | 1
    2 | 0 | 2 | 1 | 0 | 3
    3 | 1 | 1 | 0 | 0 | 2
    4 | 0 | 0 | 0 | 0 | 0
    >4 | 0 | 0 | 0 | 0 | 0
Time asleep (habitual and desired) [Mean (Standard Deviation); unit: minutes]
  Habitual | 368.0 (89.27) | 406.4 (105.29) | 371.6 (95.29) | 384.8 (78.88) | 382.6 (93.01)
  Desired | 341.7 (76.46) | 347.7 (72.05) | 331.3 (75.30) | 330.9 (64.43) | 337.8 (72.06)
Time to fall asleep (habitual and desired) [Mean (Standard Deviation); unit: minutes] — Habitual sleep time defined as the time it takes to fall asleep starting at subject's usual, later sleep time. Desired sleep time defined as the time it takes to fall asleep at subject's preferred, earlier sleep time.
  minutes
    Habitual | 83.0 (78.85) | 76.8 (59.89) | 90.4 (64.79) | 69.8 (58.72) | 80.2 (65.66)
    Desired | 167.5 (53.25) | 164.4 (51.43) | 165.0 (48.94) | 155.0 (55.61) | 163.0 (51.89)

OUTCOME MEASURES:

1. Primary Outcome: Latency to Persistent Sleep Over a 2-night Average Measured by Polysomnography (Nights 6-7)
Description: The elapsed time from the beginning of the polysomnography recording to the onset of the first 10 minutes of continuous sleep (ie, total number of epochs before the first 20 consecutive non-wake epochs divided by 2).
Time Frame: Nights 6-7
Population: Analysis was conducted on the full analysis set (FAS), which consisted of all randomized subjects who had at least a baseline assessment and 1 post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
minutes | 59.30 (6.684) | 39.40 (6.352) | 55.94 (6.482) | 55.12 (6.871)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the analysis of covariance (ANCOVA) model; Test type: Superiority or Other; p = 0.646, ANCOVA — Statistical significance was determined at the 0.05 level; Least Squares (LS) means were estimated using an ANCOVA model with treatment and pooled center as class effects and baseline value as a covariate
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.084, ANCOVA — Statistical significance was determined at the 0.05 level; LS means were estimated using an ANCOVA model with treatment and pooled center as class effects and baseline value as a covariate
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.929, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

2. Secondary Outcome: Latency to Persistent Sleep Over a 2-night Average Measured by Polysomnography (Nights 13-14)
Description: as for outcome 1
Time Frame: Nights 13-14
Population: Analysis was conducted on the FAS, which consisted of all randomized subjects who had at least a baseline assessment and 1 post-baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
minutes | 48.36 (6.849) | 38.61 (6.611) | 45.29 (6.732) | 46.64 (6.983)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.854, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.383, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.883, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

3. Secondary Outcome: Total Sleep Time Over a 2-night Average Measured by Polysomnography (Nights 6-7)
Description: The sum of all of the minutes of Stages 1, 2, 3, 4, and rapid eye movement (REM) sleep.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
minutes | 376.41 (8.158) | 383.51 (7.876) | 378.62 (8.033) | 366.23 (8.421)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.365, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.121, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.269, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

4. Secondary Outcome: Total Sleep Time Over a 2-night Average Measured by Polysomnography (Nights 13-14)
Description: The sum of all of the minutes of Stages 1, 2, 3, 4, and REM sleep.
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
minutes | 389.72 (8.866) | 378.04 (8.683) | 379.17 (8.843) | 388.51 (9.064)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.920, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.382, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.439, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

5. Secondary Outcome: Sleep Efficiency Over a 2-night Average Measured by Polysomnography (0-3 Hours) (Nights 6-7)
Description: The total sleep time divided by time-in-bed, multiplied by 100.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
percentage of time asleep | 64.49 (3.385) | 71.83 (3.213) | 65.70 (3.272) | 64.64 (3.460)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.973, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.117, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.816, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

6. Secondary Outcome: Sleep Efficiency Over a 2-night Average Measured by Polysomnography (0-3 Hours) (Nights 13-14)
Description: The total sleep time divided by time-in-bed, multiplied by 100.
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
percentage of time asleep | 69.07 (3.244) | 75.13 (3.126) | 70.19 (3.181) | 70.99 (3.286)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.661, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.341, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.853, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

7. Secondary Outcome: Sleep Efficiency Over a 2-night Average Measured by Polysomnography (0-8 Hours) (Nights 6-7)
Description: The total sleep time divided by time-in-bed, multiplied by 100.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
percentage of time asleep | 78.42 (1.701) | 79.90 (1.642) | 78.89 (1.675) | 76.30 (1.756)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.365, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.121, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.268, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

8. Secondary Outcome: Sleep Efficiency Over a 2-night Average Measured by Polysomnography (0-8 Hours) (Nights 13-14)
Description: The total sleep time divided by time-in-bed, multiplied by 100.
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
percentage of time asleep | 81.09 (1.706) | 79.33 (1.671) | 78.92 (1.702) | 80.80 (1.745)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.900, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.525, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.418, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

9. Secondary Outcome: Wake Time After Sleep Onset Over a 2-night Average Measured by Polysomnography (Nights 6-7)
Description: The number of wake minutes after the onset of persistent sleep prior to the end of recording.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
minutes | 46.26 (5.880) | 62.86 (5.704) | 51.06 (5.758) | 62.11 (6.035)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.051, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.926, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.166, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

10. Secondary Outcome: Wake Time After Sleep Onset Over a 2-night Average Measured by Polysomnography (Nights 13-14)
Description: The number of wake minutes after the onset of persistent sleep prior to the end of recording.
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
minutes | 43.36 (6.124) | 63.47 (6.032) | 59.77 (6.103) | 48.88 (6.240)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.511, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.082, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.188, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

11. Secondary Outcome: Number of Awakenings Over a 2-night Average Measured by Polysomnography (Nights 6-7)
Description: The number of times after onset of persistent sleep that there is a wake entry of at least 2 epochs in duration. Each entry must be separated by stage 2, stage 3/4 non-REM (NREM) sleep, or REM sleep to be counted.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of awakenings
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
number of awakenings | 9.22 (0.835) | 10.79 (0.795) | 10.79 (0.815) | 9.67 (0.853)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.691, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.323, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.324, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

12. Secondary Outcome: Number of Awakenings Over a 2-night Average Measured by Polysomnography (Nights 13-14)
Description: as for outcome 11
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of awakenings
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
number of awakenings | 8.08 (0.806) | 9.33 (0.783) | 9.87 (0.800) | 9.51 (0.822)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.197, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.871, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.737, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

13. Secondary Outcome: Total Wake Time Over a 2-night Average Measured by Polysomnography (Nights 6-7)
Description: The sum of all the minutes of Stage Wake from the beginning of the recording to the end of recording.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
minutes | 63.92 (6.096) | 50.67 (5.785) | 61.67 (5.892) | 63.63 (6.230)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.972, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.117, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.811, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

14. Secondary Outcome: Total Wake Time Over a 2-night Average Measured by Polysomnography (Nights 13-14)
Description: The sum of all the minutes of Stage Wake from the beginning of the recording to the end of recording.
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
minutes | 55.69 (5.841) | 44.68 (5.629) | 53.64 (5.728) | 52.19 (5.918)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.659, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.337, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.853, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

15. Secondary Outcome: Sleep Time Over a 2-night Average Measured by Polysomnography (Nights 6-7)
Description: Sleep time was measured as the clock time the subject went to sleep. Units are hours and minutes on a 24-hour clock, expressed in decimal time.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
hours on a 24-hour clock | 22.40 (0.016) | 22.36 (0.016) | 22.35 (0.016) | 22.35 (0.033)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.206, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.495, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.800, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

16. Secondary Outcome: Sleep Time Over a 2-night Average Measured by Polysomnography (Nights 13-14)
Description: as for outcome 15
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
hours on a 24-hour clock | 22.36 (0.016) | 22.36 (0.016) | 22.36 (0.016) | 22.33 (0.016)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.194, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.134, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.130, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

17. Secondary Outcome: Wake Time Over a 2-night Average Measured by Polysomnography (Nights 6-7)
Description: Wake Time was measured as the clock time that the subject got up in the morning. Units are hours and minutes on a 24-hour clock, expressed in decimal time.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 33 | 30
hours on a 24-hour clock | 06.35 (0.033) | 06.31 (0.033) | 06.30 (0.033) | 06.26 (0.033)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.063, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.156, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.521, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

18. Secondary Outcome: Wake Time Over a 2-night Average Measured by Polysomnography (Nights 13-14)
Description: as for outcome 17
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 32 | 32 | 30
hours on a 24-hour clock | 06.31 (0.066) | 06.21 (0.066) | 06.40 (0.066) | 06.26 (0.083)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.675, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.566, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.205, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

19. Secondary Outcome: Total Sleep Time Measured by Actigraphy (Nights 6-7)
Description: Total sleep time calculated using the total number of epochs (number of movements recorded by actigraphy watch worn by subject) that are less than or equal to 40, measured between the start time and end time during the nocturnal sleep interval, scored as SLEEP by the actigraphy software.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 28 | 28 | 29
minutes | 374.37 (8.741) | 393.37 (8.632) | 370.83 (8.352) | 369.05 (8.457)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.643, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.032, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.875, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

20. Secondary Outcome: Total Sleep Time Measured by Actigraphy (Nights 13-14)
Description: Total sleep time pertains to the total number of epochs (number of movements recorded by actigraphy watch worn by subject) that are less than or equal to 40, measured between the start time and end time during the nocturnal sleep interval, scored as SLEEP by the actigraphy software.
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 27 | 30 | 27
minutes | 391.61 (8.661) | 390.76 (8.982) | 370.80 (8.228) | 378.91 (8.845)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.286, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.318, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.483, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

21. Secondary Outcome: Sleep Efficiency Measured by Actigraphy (Nights 6-7)
Description: Sleep efficiency pertains to the scored total sleep time (recorded by actigraphy watch worn by subject) of the sleep interval divided by total time in bed minus total invalid time (Sleep/Wake), multiplied by 100.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 28 | 28 | 29
percentage of time asleep | 85.79 (1.117) | 83.46 (1.086) | 81.38 (1.081) | 82.72 (1.089)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.040, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.610, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.368, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

22. Secondary Outcome: Sleep Efficiency Measured by Actigraphy (Nights 13-14)
Description: as for outcome 21
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: percentage of time asleep
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 27 | 30 | 27
percentage of time asleep | 84.98 (1.349) | 82.91 (1.381) | 81.31 (1.300) | 83.24 (1.388)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.352, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.860, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.297, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

23. Secondary Outcome: Wake Time During Sleep Interval Measured by Actigraphy (Nights 6-7)
Description: Wake time during sleep is the total number of epochs (number of movements recorded by actigraphy watch worn by subject) between the start time and the end time of the given sleep interval, scored as WAKE by the software (or manually set as WAKE by the practitioner using the software), multiplied by the Epoch length in minutes.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 28 | 28 | 29
minutes | 41.81 (4.404) | 51.98 (4.298) | 54.70 (4.211) | 53.14 (4.223)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.053, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.837, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.783, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

24. Secondary Outcome: Wake Time During Sleep Interval Measured by Actigraphy (Nights 13-14)
Description: as for outcome 23
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 27 | 30 | 27
minutes | 48.11 (4.074) | 54.72 (4.185) | 52.36 (3.874) | 51.32 (4.140)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.566, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.543, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.847, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

25. Secondary Outcome: Wake Bouts Measured by Actigraphy (Nights 6-7)
Description: The number of wake bouts pertains to the total number of continuous blocks (recorded by actigraphy watch worn by subject), with one or more epochs in duration, and with each epoch of each clock scored as WAKE between the start time and the end time of the given interval.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: wake bouts
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 28 | 28 | 29
wake bouts | 20.98 (1.518) | 22.91 (1.476) | 23.32 (1.457) | 22.82 (1.442)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.356, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.964, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.799, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

26. Secondary Outcome: Wake Bouts Measured by Actigraphy (Nights 13-14)
Description: as for outcome 25
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: wake bouts
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 27 | 30 | 27
wake bouts | 23.42 (1.201) | 24.21 (1.230) | 23.52 (1.146) | 22.78 (1.206)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.698, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.385, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.641, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

27. Secondary Outcome: Sleep Latency Measured by Actigraphy (Nights 6-7)
Description: The elapsed time from the beginning of the recording to the onset of the first 10 minutes of continuous sleep (recorded by actigraphy watch worn by subject).
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 28 | 28 | 29
minutes | 12.53 (3.292) | 18.05 (3.280) | 25.00 (3.156) | 12.42 (3.129)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.979, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.194, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.004, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

28. Secondary Outcome: Sleep Latency Measured by Actigraphy (Nights 13-14)
Description: as for outcome 27
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 27 | 30 | 27
minutes | 12.10 (6.145) | 16.40 (6.460) | 25.43 (5.859) | 12.36 (6.169)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.975, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.639, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.109, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

29. Secondary Outcome: Sleep Time Measured by Actigraphy (Nights 6-7)
Description: Clock time subject goes to sleep (recorded by actigraphy watch worn by subject). Units are hours and minutes on a 24-hour clock, expressed in decimal time.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 28 | 28 | 29
hours on a 24-hour clock | 23.28 (0.150) | 22.75 (0.150) | 23.11 (0.150) | 23.31 (0.150)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.823, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.004, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.296, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

30. Secondary Outcome: Sleep Time Measured by Actigraphy (Nights 13-14)
Description: as for outcome 29
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 27 | 30 | 27
hours on a 24-hour clock | 22.83 (0.150) | 22.71 (0.166) | 23.11 (0.150) | 23.18 (0.150)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.092, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.025, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.732, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

31. Secondary Outcome: Wake Time Measured by Actigraphy (Nights 6-7)
Description: Clock time subject wakes up (recorded by actigraphy watch worn by subject). Units are hours and minutes on a 24-hour clock, expressed in decimal time.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 28 | 28 | 29
hours on a 24-hour clock | 06.20 (0.116) | 06.18 (0.116) | 06.23 (0.116) | 06.36 (0.116)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.298, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.276, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.430, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

32. Secondary Outcome: Wake Time Measured by Actigraphy (Nights 13-14)
Description: as for outcome 31
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 26 | 27 | 30 | 27
hours on a 24-hour clock | 06.13 (0.133) | 06.08 (0.133) | 06.16 (0.133) | 06.30 (0.133)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.349, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.203, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.444, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

33. Secondary Outcome: Subjective Sleep Latency Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: Subjective sleep latency was an average of 2 nights responses and measured by post-sleep questionnaire in response to the question, "How long do you think it took you to fall asleep last night?"
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 34 | 30
minutes | 103.55 (8.301) | 84.46 (8.087) | 92.79 (7.930) | 97.28 (8.491)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.581, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.257, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.688, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

34. Secondary Outcome: Subjective Sleep Latency Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 33
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 28 | 29 | 32 | 30
minutes | 80.57 (7.406) | 69.40 (7.423) | 77.29 (7.178) | 74.75 (7.407)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.561, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.595, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.795, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

35. Secondary Outcome: Subjective Total Sleep Time Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: Subjective total sleep time was an average of 2 nights responses and measured by post-sleep questionnaire in response to the question, "How long (total hours and minutes) do you think you slept last night?"
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 34 | 30
minutes | 348.10 (10.302) | 370.14 (10.067) | 360.57 (9.883) | 341.76 (10.571)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.655, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.177, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.044, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

36. Secondary Outcome: Subjective Total Sleep Time Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 35
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 28 | 29 | 32 | 30
minutes | 379.20 (10.490) | 375.73 (10.532) | 365.14 (10.229) | 368.99 (10.513)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.475, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.635, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.782, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

37. Secondary Outcome: Subjective Wake Time After Sleep Onset Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: Subjective wake time after sleep onset was an average of 2 nights responses and measured by post-sleep questionnaire in response to the question, "Did you wake up during the night? If "yes", what is the total time you think you were awake?"
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 34 | 30
minutes | 35.15 (7.084) | 52.52 (6.671) | 34.41 (6.659) | 47.84 (7.100)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.192, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.618, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.152, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

38. Secondary Outcome: Subjective Wake Time After Sleep Onset Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 37
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 28 | 29 | 32 | 30
minutes | 23.49 (5.882) | 45.54 (5.877) | 28.66 (5.669) | 30.52 (5.794)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.379, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.057, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.808, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

39. Secondary Outcome: Subjective Number of Awakenings Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: Subjective number of awakenings was an average of 2 nights responses and measured by post-sleep questionnaire in response to the question, "Did you wake up during the night? If "yes", how many times do you think you woke up?"
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of awakenings
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 25 | 27 | 21 | 22
number of awakenings | 2.68 (0.364) | 3.72 (0.382) | 2.92 (0.385) | 3.23 (0.383)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.284, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.344, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.558, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

40. Secondary Outcome: Subjective Number of Awakenings Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 39
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: number of awakenings
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 19 | 22 | 21 | 22
number of awakenings | 2.94 (0.456) | 3.72 (0.427) | 3.33 (0.443) | 3.04 (0.423)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.867, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.244, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.620, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

41. Secondary Outcome: Subjective Sleep Quality Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: Subjective sleep quality was an average of 2 nights responses and measured by post-sleep questionnaire in response to the question, "How would you describe the quality of your sleep last night?" Scores were based on the following scale: Extremely Poor=7; Very Poor=6; Poor=5; Fair=4; Good=3; Very Good=2; Excellent=1.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 34 | 30
scores on a scale | 4.45 (0.169) | 4.61 (0.166) | 4.33 (0.162) | 4.74 (0.173)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.206, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.559, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.074, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

42. Secondary Outcome: Subjective Sleep Quality Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 41
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 28 | 29 | 32 | 30
scores on a scale | 4.27 (0.184) | 4.35 (0.185) | 4.03 (0.179) | 4.20 (0.184)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.796, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.546, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.479, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

43. Secondary Outcome: Subjective Sleep Time Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: Subjective sleep time was an average of 2 nights responses and measured by post-sleep questionnaire in response to the question, "What time did you try to go to sleep last night?" Units are hours and minutes on a 24-hour clock, expressed in decimal time.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 34 | 30
hours on a 24-hour clock | 10.36 (0.066) | 10.41 (0.066) | 10.40 (0.066) | 10.40 (0.066)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.766, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.912, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.952, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

44. Secondary Outcome: Subjective Sleep Time Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 43
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 28 | 29 | 32 | 30
hours on a 24-hour clock | 10.36 (0.066) | 10.30 (0.066) | 10.36 (0.066) | 10.40 (0.066)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.722, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.262, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.717, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

45. Secondary Outcome: Subjective Getting up in the Morning Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: The score was an average of 2 nights responses. If subjects had a work or school day, the answer to, "How easy was it for you to wake or get up in the morning when on a school or working night?" was based on the following scale: Extremely Difficult =7; Very Difficult =6; Difficult =5; Neither =4; Easy =3; Very Easy =2; Extremely Easy =1.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 25 | 29 | 31 | 24
scores on a scale | 4.68 (0.224) | 4.76 (0.202) | 4.67 (0.178) | 4.88 (0.203)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.498, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.664, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.428, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

46. Secondary Outcome: Subjective Getting up in the Morning Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 45
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 24 | 23 | 26 | 25
scores on a scale | 4.46 (0.219) | 4.66 (0.217) | 4.30 (0.191) | 4.28 (0.198)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.519, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.179, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.935, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

47. Secondary Outcome: Subjective Ability to Concentrate in the Morning Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: Subjective ability to concentrate was an average of 2 nights responses and measured by post-sleep questionnaire in response to the question, "How would you describe your ability to concentrate this morning?" Scores were based on the following scale: Extremely Poor=7; Very Poor=6; Poor=5; Fair=4; Good=3; Very Good=2; Excellent=1.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 33 | 34 | 30
scores on a scale | 4.31 (0.155) | 4.30 (0.151) | 4.40 (0.148) | 4.48 (0.159)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.425, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.406, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.720, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

48. Secondary Outcome: Subjective Ability to Concentrate in the Morning Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 47
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 28 | 29 | 32 | 30
scores on a scale | 3.77 (0.164) | 4.17 (0.164) | 4.01 (0.159) | 4.01 (0.164)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.294, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.474, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.999, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

49. Secondary Outcome: Subjective Level of Alertness Measured by a Post-sleep Questionnaire (Nights 6-7)
Description: Subjective level of alertness was an average of 2 nights responses and measured by post-sleep questionnaire in response to the question, "How would you describe your level of alertness this morning?" Scores were based on the following scale: Extremely Poor=7; Very Poor=6; Poor=5; Fair=4; Good=3; Very Good=2; Excellent=1.
Time Frame: Nights 6-7
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 31 | 31 | 34 | 30
scores on a scale | 4.43 (0.158) | 4.32 (0.155) | 4.33 (0.152) | 4.53 (0.163)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.655, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.331, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.362, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

50. Secondary Outcome: Subjective Level of Alertness Measured by a Post-sleep Questionnaire (Nights 13-14)
Description: as for outcome 49
Time Frame: Nights 13-14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 28 | 29 | 32 | 30
scores on a scale | 4.02 (0.181) | 4.32 (0.181) | 3.99 (0.176) | 4.12 (0.182)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.684, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.399, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.611, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

51. Secondary Outcome: Next Morning Residual Effects Assessments of Psychomotor and Cognitive Function Via Digit Symbol Substitution Test
Description: The number of correct digit-for-number substitutions on a Digit Symbol Substitution Test in the 90-second period was recorded to assess psychomotor and cognitive function. The score was the average of 2 mornings' tests. Worst Value: 0. Best Value: No Limit.
Time Frame: Day 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 31 | 32 | 29
Scores on a scale | 44.1 (1.77) | 42.4 (1.74) | 39.9 (1.74) | 40.6 (1.83)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.157, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.463, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.774, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

52. Secondary Outcome: Next Morning Residual Effects Assessments of Psychomotor and Cognitive Function Via Memory Recall Test--Immediate
Description: After 16 words were read to a subject, a subject was given 2 minutes to write down as many words as he/she remembered. The correct number of words written was scored, and the average of 2 mornings' tests was calculated.
Time Frame: Day 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 30 | 32 | 29
score | 8.1 (0.39) | 7.7 (0.40) | 8.6 (0.39) | 8.6 (0.41)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.413, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.093, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.982, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

53. Secondary Outcome: Next Morning Residual Effects Assessments of Psychomotor and Cognitive Function Via Memory Recall Test--Delayed
Description: After 16 words were read to a subject, a subject waited 1 minute and then was given 2 minutes to write down as many words as he/she remembered. The correct number of words written was scored, and the average of 2 mornings' tests was calculated.
Time Frame: Day 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 30 | 32 | 29
score | 6.5 (0.51) | 5.9 (0.51) | 6.7 (0.50) | 7.1 (0.52)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.441, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.082, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.549, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

54. Secondary Outcome: Visual Analogue Scale for Mood
Description: Subjects marked visual scales (in millimeters) that represented ranges of emotions (eg, calm to anxious; normal to bloated; energetic to fatigued). Individual subject composite scores were calculated, and the average of 2 tests were analyzed. Worst Value: 0 mm. Best Value: 100 mm. The farther to the left a subject marks, the better their mood; farther to the right, the more distressed the mood. Higher numbers indicate a more distressed mood.
Time Frame: Day 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 31 | 32 | 29
Units on a scale | 34.2 (3.20) | 33.4 (3.15) | 34.3 (3.17) | 33.4 (3.31)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.860, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.997, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.834, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

55. Secondary Outcome: Visual Analogue Scale for Feelings
Description: Subjects marked visual scales (in millimeters) that represented ranges of emotions (eg, calm to anxious; normal to bloated; energetic to fatigued). Individual subject composite scores were calculated, and the average of 2 tests were analyzed. Worst Value:0 mm.. Best Value:100 mm.. The farther to the left a subject marks, the better their mood; farther to the right, the more distressed the mood. Higher numbers indicate a more distressed mood.
Time Frame: Day 15
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 30 | 31 | 32 | 30
Units on a scale | 37.3 (1.52) | 34.8 (1.50) | 36.8 (1.50) | 36.9 (1.57)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.837, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.321, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.978, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

56. Secondary Outcome: The Time of Dim Light Melatonin Secretion Onset
Description: Linear Dim Light Melatonin Secretion Onset is defined as the first time of the evening (on a 24-hour clock) when the melatonin level rises above 3.0 pg/ml with a positive slope. Units are hours and minutes on a 24-hour clock, expressed in decimal time.
Time Frame: Day 15
Population: The melatonin set included all subjects who had saliva samples collected under dim light conditions for melatonin measurement.
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 25 | 29 | 31 | 25
hours on a 24-hour clock | 21.40 (0.183) | 21.30 (0.166) | 20.93 (0.166) | 21.21 (0.200)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.513, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.751, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.242, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

57. Secondary Outcome: The Time of Dim Light Melatonin Secretion Offset
Description: Dim Light Melatonin Secretion Offset is defined as the first time of the morning (on a 24-hour clock) when the melatonin drops to below 3 pg/mL with a negative slope. Units are hours and minutes on a 24-hour clock, expressed in decimal time.
Time Frame: Day 15
Population: as for outcome 56
Measure: Least Squares Mean (Standard Error); unit: hours on a 24-hour clock
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 25 | 29 | 31 | 25
hours on a 24-hour clock | 11.21 (0.250) | 10.73 (0.250) | 10.96 (0.250) | 10.85 (0.283)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.307, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.765, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.727, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

58. Secondary Outcome: The Total Duration of Secretion of Melatonin
Description: The total duration of time from Dim Light Melatonin Secretion Onset to Dim Light Melatonin Secretion Offset.
Time Frame: Day 15
Population: as for outcome 56
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 25 | 29 | 31 | 25
minutes | 1021.8 (34.13) | 1003.1 (31.98) | 980.2 (31.43) | 1027.9 (36.39)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.902, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.590, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.290, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

59. Secondary Outcome: The Area Under the Concentration-time Curve of Melatonin From 0 to 24 Hours
Description: Area under the concentration-time curve is a measure of total drug exposure.
Time Frame: Day 15
Population: as for outcome 56
Measure: Least Squares Mean (Standard Error); unit: μg/dL/hour
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 25 | 29 | 31 | 25
μg/dL/hour | 608.5 (40.13) | 563.3 (38.08) | 528.3 (37.35) | 631.5 (42.77)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.685, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.214, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.055, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

60. Secondary Outcome: Average Cmax (Maximum Observed Plasma Concentration) Calculated as the Average of Three Highest Cmax Observations Within the Sampling Period.
Description: Average Cmax calculated as the average of three highest Cmax observations within the sampling period.
Time Frame: Day 15
Population: as for outcome 56
Measure: Least Squares Mean (Standard Error); unit: μg/dL
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Number analyzed (Participants) | 25 | 29 | 31 | 25
μg/dL | 75.3 (5.12) | 69.3 (4.84) | 65.2 (4.77) | 79.2 (5.46)
Statistical Analysis 1: Comparison: Ramelteon 1 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.589, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Ramelteon 4 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.156, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Ramelteon 8 mg QD vs Placebo QD; The comparison between the 2 treatment groups was made using the ANCOVA model; Test type: Superiority or Other; p = 0.041, ANCOVA — Statistical significance was determined at the 0.05 level; [statistical method as in outcome 1, analysis 2]

ADVERSE EVENTS:
Description: There were no Serious Adverse Events
Arm/Group | Ramelteon 1 mg QD | Ramelteon 4 mg QD | Ramelteon 8 mg QD | Placebo QD
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33 | 0/35 | 0/32
Other Adverse Events (participants affected / at risk) | 7/32 | 5/33 | 6/35 | 4/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ramelteon 1 mg QD (N=32) | Ramelteon 4 mg QD (N=33) | Ramelteon 8 mg QD (N=35) | Placebo QD (N=32)
Blood Creatine Phosphokinase Increased (Investigations) | 1 | 0 | 2 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 1 | 3 | 1
Somnolence (Nervous system disorders) | 2 | 2 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release; such communications can be embargoed for a period up to 150 days to permit actions necessary to preserve sponsor's intellectual property. Sponsor can request changes to the results communication only for the purpose of removing non study related information that is proprietary and confidential to sponsor. Sponsor can require delay of a results communication until the study has been completed at all participating sites.